CLINICAL TRIAL: NCT06583109
Title: Establishment and Application of Prediction Model of Treatment Efficacy for Age-related Macular Degeneration Based on Multi-source Imaging Modalities
Brief Title: Prediction Model of Treatment Efficacy for Age-related Macular Degeneration Based on Multi-source Imaging Modalities
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: BJ-2024-089
Record Dates: First submitted 2024-09-01; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-09

CONDITIONS: Age-related Macular Degeneration (ARMD)
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
Age-related macular degeneration (AMD) is one of the main causes of blindness in the elderly population. Intraocular injection of anti-VEGF drugs for neovascular AMD (nAMD) is the main treatment method at present. However, patients have different responses to anti-VEGF therapy, and some patients do not respond well to short - and long-term treatment.

In this study, a retrospective study was adopted to collate and analyze the clinical data and imaging data of nAMD in the past, and to extract the imaging features from the multimodal modalities before and after treatment for deep learning, and to evaluate and quantify the clinical features, and to construct two multi-source feature models for predicting the short-term and long-term prognosis of nAMD patients. By verifying the accuracy of the model to predict the curative effect, the classification efficiency of the above characteristic models was compared, and the optimal model was selected. Its clinical application value was evaluated by calibration curve and decision curve. In addition, patients with poor treatment response in the study cohort were retrospectively analyzed, and the efficacy and safety of the combination of other treatment options in the actual clinic were analyzed. The purpose of this study is to provide scientific basis for early prediction, dynamic monitoring and optimization of overall treatment strategies for nAMD.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with nAMD by ophthalmic examinations including OCT, OCTA, FFA and ICGA;
* Complete clinical data and imaging data of patients were available at baseline, 3 months and 1 year after anti-VEGF treatment.

Exclusion Criteria:

* Medical records showed other diseases affecting visual function or fundus imaging, such as macular edema, glaucoma, ocular trauma, etc;
* Medical records showed that two or more macular lesions coexist in the affected eye;
* Medical records showed that patients received other treatments within 1 year of anti-VEGF therapy, such as intraocular laser therapy or ocular surgery;
* Medical records showed that there were ocular media opacity, dense macular hemorrhage, or severe macular atrophy, resulting in the inability to accurately measure the required parameters;
* Medical records showed the use of drugs known to cause retinal toxicity, or a history of radiation exposure.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with nAMD who had completed routine follow-up within 1 year after standard anti-VEGF therapy with complete demographic and ophthalmological data were retrospectively collected.
Sampling Method: Non-Probability Sample
Enrollment: 2600 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
BCVA | Baseline, 3 months after anti-VEGF treatment, 1 year after anti-VEGF treatment
  best-corrected visual acuity using LogMAR

SECONDARY OUTCOMES:
CMT | Baseline, 3 months after anti-VEGF treatment, 1 year after anti-VEGF treatment
  central macular thickness measured on OCT

IPD SHARING:
Plan to Share IPD: No